CLINICAL TRIAL: NCT01270438
Title: A Phase 2 Study of RO4929097 (NSC 749225) in Combination With FOLFOX Plus Bevacizumab Versus FOLFOX Plus Bevacizumab Alone for the First-Line Treatment of Patients With Metastatic Colorectal Cancer (NCI #8467)
Brief Title: Combination Chemotherapy and Bevacizumab With or Without RO4929097 in Treating Patients With Metastatic Colorectal Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02571; NCI-2011-02571 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000692198; MSKCC-10191; 10-191 (Other: Memorial Sloan Kettering Cancer Center); 8467 (Other: CTEP); U01CA069856 (NIH); N01CM62206 (NIH)
Record Dates: First submitted 2011-01-04; First posted 2011-01-05 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Adenocarcinoma of the Colon; Adenocarcinoma of the Rectum; Recurrent Colon Cancer; Recurrent Rectal Cancer; Stage IVA Colon Cancer; Stage IVA Rectal Cancer; Stage IVB Colon Cancer; Stage IVB Rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms; Rectal Neoplasms | interventions — Folfox protocol; 2,2-dimethyl-N-(6-oxo-6,7-dihydro-5H-dibenzo(b,d)azepin-7-yl)-N'-(2,2,3,3,3-pentafluoropropyl)malonamide; Bevacizumab; Oxaliplatin; Leucovorin; Fluorouracil

ARMS (2):
- Arm I (RO4929097, combination chemotherapy, bevacizumab) (Experimental): Patients receive FOLFOX6 regimen comprising oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, fluorouracil IV continuously over 46 hours, and bevacizumab IV over 30-90 minutes on days 1-2. Patients also receive oral gamma-secretase inhibitor RO4929097 on days 1-3 and 8-10. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: FOLFOX regimen; Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097; Biological: bevacizumab; Drug: oxaliplatin; Drug: leucovorin calcium; Drug: fluorouracil
- Arm II (combination chemotherapy, bevacizumab) (Experimental): Patients receive FOLFOX6 regimen and bevacizumab as in arm I. Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: FOLFOX regimen; Biological: bevacizumab; Drug: oxaliplatin; Drug: leucovorin calcium; Drug: fluorouracil

INTERVENTIONS:
Drug: FOLFOX regimen — Given IV
Drug: gamma-secretase/Notch signalling pathway inhibitor RO4929097 — Given orally
  Arms: Arm I (RO4929097, combination chemotherapy, bevacizumab)
Biological: bevacizumab — Given IV
Drug: oxaliplatin — Given IV
Drug: leucovorin calcium — Given IV
Drug: fluorouracil — Given IV

SUMMARY:
This phase II clinical trial is studying how well giving combination chemotherapy and bevacizumab with or without RO4929097 works in treating patients with metastatic colorectal cancer. Drugs used in chemotherapy, such as oxaliplatin, leucovorin calcium, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. RO4929097 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether combination chemotherapy and bevacizumab is more effective with RO4929097 in treating patients with colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the efficacy, as determined by progression-free survival, of FOLFOX6 and bevacizumab with versus without gamma-secretase inhibitor RO4929097 (RO4929097).

SECONDARY OBJECTIVES:

I. To estimate the clinical benefit of RO4929097 in combination with mFOLFOX6 and bevacizumab, as measured by objective response rate.

II. To evaluate the safety and tolerability of RO4929097 in combination with mFOLFOX6 chemotherapy and bevacizumab.

III. To evaluate the pharmacokinetics (PK) and pharmacodynamics (PD) of RO4929097 in combination with mFOLFOX6 and bevacizumab.

IV. To investigate PD response of RO4929097 in combination with mFOLFOX6 chemotherapy and bevacizumab, as assessed by direct measurement of gamma-secretase enzyme activity, in tumor samples.

V. (Exploratory) To investigate the Notch signaling pathway genes targeted by RO4929097 in combination with mFOLFOX6 chemotherapy and bevacizumab and correlate with clinical outcome.

VI. (Exploratory) To investigate the Ras signaling pathway genes targeted by RO4929097 in combination with mFOLFOX6 chemotherapy and bevacizumab and correlate with clinical outcome.

VII. (Exploratory) To investigate putative colorectal cancer stem cells targeted by RO4929097 in combination with mFOLFOX6 chemotherapy and bevacizumab and correlate with clinical outcome.

OUTLINE: This is a multicenter study. Patients are stratified according to participating center, prior therapy (adjuvant/neoadjuvant vs none), and number of organs* involved by metastases (1 vs > 1). Patients are randomized to 1 of 2 treatment arms.

NOTE: *Lesions all in the liver would be considered as 1 organ involved.

ARM I: Patients receive FOLFOX6 regimen comprising oxaliplatin intravenously (IV) over 2 hours, leucovorin calcium IV over 2 hours, fluorouracil IV continuously over 46 hours, and bevacizumab IV over 30-90 minutes on days 1-2. Patients also receive oral gamma-secretase inhibitor RO4929097 on days 1-3 and 8-10.

Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity (RO4929097 is given for up to 12 courses).

ARM II: Patients receive FOLFOX6 regimen and bevacizumab as in arm I.

Courses repeat every 14 days in the absence of disease progression or unacceptable toxicity. Patients may undergo blood sample collection at baseline and periodically during study for pharmacokinetic, pharmacodynamic, and correlative studies.

After completion of study therapy, patients are followed up for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the colon or adenocarcinoma of the rectum

  * Metastatic disease by imaging
* Measurable disease, defined as ≥ 1 lesion that can be accurately measured in ≥ 1 dimension (longest diameter to be recorded) as ≥ 20mm by conventional techniques or as ≥ 10 mm by spiral CT scan
* No known brain metastases
* ECOG performance status 0-1
* ANC ≥ 1,500/mm³
* WBC ≥ 3,000/mm³
* Platelet count ≥ 100,000/mm³ (without a platelet transfusion ≤ 14 days prior to study)
* Hemoglobin ≥ 9 g/dL
* Serum creatinine ≤ 1.5 times upper limit of normal (ULN)
* Urine protein:creatinine ≤ 0.5 or proteinuria < 1,000 mg on 24-hour urine collection
* Total bilirubin ≤ 1.5 times ULN
* AST and ALT ≤ 2.5 times ULN (≤ 5.0 times ULN for patients with liver metastases)
* Albumin ≥ 2.5 g/dL
* Amylase ≤ 2 times ULN
* Lipase ≤ 2 times ULN
* PTT ≤ 1.2 times ULN
* INR ≤ 1.2 times ULN
* No patients with uncontrolled hypophosphatemia, hypocalcemia, hypomagnesemia, hyponatremia, or hypokalemia defined as less than the lower limit of normal for the institution, despite adequateelectrolyte supplementation
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use two forms of contraception (i.e., barrier contraception and one other method of contraception) prior to, during, and for ≥ 12 months after study participation
* Patients must not have current evidence of or history of another malignancy except adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other curatively treated solid tumors with no evidence of disease for ≥ 3 years prior to enrollment
* Able to swallow capsules
* No malabsorption syndrome or other condition that would interfere with intestinal absorption
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to gamma-secretase inhibitor RO4929097 used in the study
* No clinically important history of liver disease, including known viral, other hepatitis, or cirrhosis
* No uncontrolled intercurrent illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * A history of torsades de pointes or other significant cardiac arrhythmias
  * Psychiatric illness and/or social situations that would limit compliance with study requirements
* No baseline QTcF > 450 msec (male) or QTcF > 470msec (female)
* No serious or non-healing wound, ulcer, or bone fracture
* No history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the past 6 months
* No significant traumatic injury within the past 28 days
* No clinically significant cardiovascular disease, including any of the following:

  * Inadequately controlled hypertension (systolic BP > 160 mm Hg and/or diastolic BP > 90 mm Hg despite antihypertension medication)
  * History of cerebrovascular accident within the past 6 months
  * Myocardial infarction or unstable angina within the past 6 months
  * NYHA grade II-IV congestive heart failure
  * Serious and inadequately controlled cardiac arrhythmia
* No requirement for antiarrhythmics or other medications known to prolong QTc
* No significant vascular disease (e.g., aortic aneurysm, requiring surgical repair, history of aortic dissection, or recent peripheral arterial thrombosis) within the past 6 months
* No clinically significant peripheral vascular disease
* No evidence of bleeding diathesis or coagulopathy
* No known hypersensitivity to Chinese hamster ovary cell products or other recombinant human antibodies
* Recovered to < NCI CTCAE grade 2 toxicities related to prior therapy
* No prior adjuvant or neoadjuvant chemotherapy for colorectal cancers within 12 months of development of metastases
* No prior chemotherapy or gamma-secretase inhibitors or other investigational agents for metastatic colorectal cancer
* No prior radiotherapy for colorectal cancers including in the neoadjuvant or adjuvant setting within 12 months of development of metastases
* No major surgical procedure or open biopsy within the past 28 days and no anticipation of need for major surgical procedures during the course of the study
* No concurrent medications with narrow therapeutic indices that are metabolized by cytochrome P450 (CYP450), including warfarin sodium (Coumadin®)

  * Patients who switch from warfarin sodium to alternative anti-coagulant agents allowed
* No concurrent medications that are strong inducers, inhibitors, or substrates of CYP3A4, including ketoconazole and grapefruit juice
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-12 (Actual); Primary Completion 2011-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Progression-free survival of patients treated with FOLFOX6 plus bevacizumab with or without gamma-secretase inhibitor RO4929097 | From start of treatment to time of progression, assessed up to 12 months
  Progression is defined as changes in RECIST 1.1-defined imaging, progression in non-target lesions as defined by RECIST 1.1, unequivocal clinical deterioration, or death from any cause.

SECONDARY OUTCOMES:
Objective response rate (complete or partial response) as measured by RECIST | Assessed up to 12 months
  Estimated using the binomial distribution and exact 95% confidence intervals (CI) will be provided.
Incidence of dose-limiting and non-dose-limiting toxicities | Assessed up to 12 months
  Summarized using descriptive statistics.
Pharmacokinetics and pharmacodynamics of gamma-secretase inhibitor RO4929097 | Baseline, and day 1 of courses 1 and 2
  Computed using non- compartmental methods for RO4929097 and will be correlated with clinical parameters using Cox regression model for association with survival and PFS and Wilcoxon rank sum test for response.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Segal, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (3):
- United States (3):
  - Mayo Clinic, Rochester, Minnesota
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio